CLINICAL TRIAL: NCT02847884
Title: IDeaL Pilot Study - Infliximab Dose to Level: Pilot Study
Acronym: IDeaL
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: The Hospital for Sick Children (Other); The Children's Hospital of Winnipeg (Other); Alberta Children's Hospital (Other); Provincial Health Services Authority British Columbia (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: UAlberta; Pro00056259 (Other: University of Alberta HREB Number)
Record Dates: First submitted 2015-11-30; First posted 2016-07-28 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2017-11

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease
Keywords: IBD; Crohn's disease; Remicade; Infliximab; Level; Drug Level; Children
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected to determine IFX levels and serum cytokines. Stool will be collected for calprotectin. Urine will be collected for metabolomics.
  If a child undergoes endoscopy or surgery during the 8 weeks after beginning IFX, a specimen will be collected for tissue cytokine assay.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Infliximab — Patients will be prescribed Infliximab as a standard of care regardless of study participation.
  Other Names: Remicade

SUMMARY:
Crohn's disease (CD) is a lifelong condition of inflammation in the bowel. CD can affect any part of the gastrointestinal tract from mouth to anus. Symptoms can include: tiredness, stomach pain, diarrhea (which may be bloody if the disease is severe), fever, weight loss, skin rashes, arthritis and inflammation of the eye.

Infliximab-IFX (Remicade®) is a medication that is used to treat CD in adults and children. In adults it has been shown that the amount of this drug a person has in their blood can show how well it is working for them. Health Canada has approved Infliximab -IFX for the treatment of CD in children 9 and older. In Canada, doctors may prescribe Inflixmab to younger children when other therapies do not resolve their disease symptoms. This is called "off-label" use of Infliximab.

IFX levels in the body and consequently its efficacy can be influenced by many biological characteristics within the patient's body. In about 17% of those treated with IFX, the patient's immune response against IFX may lead to a three to fivefold increased risk of loss of response. This immune response to the medication often occurs when drug levels are undetectable in the body. Thus it is in order to achieve best results with this treatment, physicians need to be able to adjust dosing specific to each patient. A recent study has shown that 29% of children have an undetectable IFX level at the 4th medication infusion. Up to 40% of patients receiving scheduled IFX have undetectable drug level prior to their next infusion.

In order to minimize the loss of response, we hope to conduct an observational cohort study of pediatric patients treated with IFX.

This open label, cohort study aims to:

1. Determine the pharmacokinetics of IFX in children with CD and the factors that affect IFX levels during the first three loading infusions
2. Obtain data to create a model that can guide and adjust the IFX dose and frequency to achieve optimal trough level between 5 and 10 ug /ml at 14 weeks.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory bowel disease characterized by inflammation that can affect any part of the gastrointestinal tract from mouth to anus. Other complications may occur outside the gastrointestinal tract and include: anemia, skin rashes, arthritis, inflammation of the eye, and tiredness. Symptoms often include: abdominal pain, diarrhea (which may be bloody if inflammation is severe), fever and weight loss. Crohn's disease is caused by a combination of environmental, immune and bacterial factors in genetically susceptible individuals. It results in a chronic inflammatory disorder, in which the body's immune system attacks the gastrointestinal tract possibly directed at microbial antigens. The estimated prevalence of CD in Canada is 234 per 100,000 persons, with an incidence rate of 13.4 per 100,000. There are no medications or surgical procedures that can cure Crohn's disease. Treatment options help with symptoms, maintain remission, and prevent relapse. The burden of disease is high with disease flares and complications leading to hospitalizations, surgeries, school and work absenteeism, and impaired quality of life.

Infliximab (IFX) is a murine chimeric lgGl anti-TNFa monoclonal antibody shown in landmark clinical trials to be well-tolerated and effective for induction, and maintenance, of remission in pediatric and adult CD and ulcerative colitis. In Canada, the safety and efficacy of IFX is not established in children under the age of 9, yet is often prescribed to younger children off label when other therapies do not resolve their disease symptoms. IFX can be influenced by multiple factors such as body mass index (BMI), serum albumin level, burden of inflammation and the concomitant use of immunosuppressive medications. Loss of response to IFX can either be a result of Antibodies to IFX (ATI) or insufficient serum IFX level.

ATI have been shown to develop in about 17% of those treated with IFX. The risk for development of ATI is even higher in those who receive IFX mono-therapy, compared to those receiving concomitant immunomodulator. It is now clear that those with persistent ATI have a three to fivefold increased risk of loss of response to IFX compared to those without ATI. ATI appears to interfere with the bioactivity of IFX and those patients who develop ATI are more likely to subsequently manifest infusion reactions, including anaphylaxis.

The standard infusion regimen for IFX is three loading dose of 5mg/kg (dose is often rounded up to the nearest 100mg) at 0, 2, 6 weeks then every 8 weeks thereafter. The trough level of IFX after the 3rd loading dose (week 14 - i.e. before the 4th infusion) is often found to be at greatest risk of being low; especially in children.

A recent study has shown that 29% of children have an undetectable IFX level at the 4th medication infusion. A trough level of 5 ug /ml at this time point is associated with higher remission rates. Conversely, a low trough level (< 2.2 ug/ml) at week 14 predicts IFX discontinuation. Up to 40% of patients receiving scheduled IFX have undetectable drug level prior to their next infusion. However, whether having undetectable IFX level at trough increases the risk of ATI formation is currently unclear. Moreover, it is unknown if dosing adjustments based on trough levels will change rates of antibody formation to IFX and the sustained efficacy of IFX nor how we can achieve desired serum levels at clinically relevant time-points, mainly because the pharmacokinetics of IFX in children has not been well studied.

Most trials assessing IFX trough levels and ATI have been performed retrospectively. A recent meta-analysis of the impact of ATI and IFX level in IBD showed that the presence of ATI is associated with a significantly higher risk of loss of clinical response to IFX and lower serum IFX levels in patients with IBD. One prospective trial of 270 adult IBD patients who were in remission on IFX maintenance therapy had their regimen modified to achieve trough IFX level between 3-7 ug/ml, and were then randomized to further dosing and optimization adjustments based on IFX trough levels - level-based (LB) - or on clinical symptoms (CB}. The primary endpoint of remission after 1 year was similar at 70%. ATI was 0 with LB and 2.7% with CB. However, 17% of CB required rescue therapy with either corticosteroids, increased doses of IFX or a switch to another Anti-TNFa (Vande Casteele UEGW 2013 Abstract). There are currently no prospective studies in pediatric patients to assess a treat-to-level of IFX strategy in Crohn's disease.

Several authors have suggested that a median trough level of > 3 ug/ml (range 2.3 to 4.9) is associated with maintenance of remission. However this value tends to reflect the limit of detection of the assay used rather than the actual biologic threshold. Lamblin reported a higher IFX level of 6.33ug /ml to be associated with higher remission rates compared to a level of 3.39 ug /ml. Based on these authors' modeling, a level 5.6 ug /ml would lead to lower inflammatory burden based on C reactive protein (CRP} < 5 ug /ml. In the most recent largest retrospective study on IFX in Inflammatory Bowel Disease (IBD) patients (n=l36}, Arias reported that a level of 7.9 ug /ml gave a 57% sensitivity and 80% specificity for predicting best sustained response to IFX. Based on the above data we hypothesize that the ideal trough level is likely between 5 and 10 ug /ml. The upper range of this trough level range is very close to the upper interquartile range in the Arias' study.

A further barrier to knowledge advancement emanates from recent changes in laboratory techniques used to assess serum IFX levels and ATI. A private laboratory in the United States, Prometheus, had previously been the only accessible laboratory where clinicians could obtain serum IFX and ATI levels using an enzyme-linked immuno sorbent assay (ELISA). Recently, they stopped performing the ELISA test and moved to an extremely expensive homogeneous mobility shift assay (HMSA) for the measurement of IFX and ATI. The advantage of this new test is the ability to detect the presence of ATI and IFX in the serum at the same time. With the previous ELISA test, ATI were not measurable in the presence of IFX, thus ATI status was typically labeled as "inconclusive" in this setting. Despite these advantages, there is currently no evidence to justify the use more sensitive but expensive HMSA test in the clinical setting and in particular there is no supporting evidence to warrant the use of this test as part of treat to level strategy.

At a time when therapeutic drug monitoring of IFX and precision dosing of biologic agents are becoming increasingly hot topics, Alberta Health Services has refused to pay for HMSA testing in patients treated with IFX because of the exorbitant costs. In an attempt to overcome this barrier to precision care, the biochemistry laboratory at the University Hospital (UAH), under the leadership of Dr Connie Prosser, has developed a locally developed (ELISA) for IFX level and ATI at a fraction of the cost charged by Prometheus ($50 for IFX level and $50 for ATI- total $100 for both tests compared to US $2500 for both IFX and ATI per test). The UAH test has been validated in a local study and was able to measure the IFX level down to 0.4 ug/ml, with very good inter- and intra- assay precision. Based on patient samples, the correlation between the UAH test and the HMSA results is excellent (R2= 0.92 for values ranging from <0.4 ug/ml to >45 ug/ml and R2 = 0.98 for values <20 ug/ml). ATI (unbound) can be measured at levels ≥ 2 ug/ml in samples having an IFX concentration < 10 ug/ml. A second ELISA is available which measures total ATI (i.e. free and bound to circulating IFX), and can detect antibody in samples with higher IFX concentrations if needed. This test is now available for clinical use in the Edmonton Zone. However the current indication for the test is only for those patients who exhibit clinical loss of response to IFX. Dose Optimization is common, 70% of us dose optimize clinically. Early dose optimization after third infusion likely to be better. How to dose optimize is unclear.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent form by the participant's parent or legal guardian, where applicable assent from the participant must also be obtained.
* Aged 2 to 17 years of age
* Known diagnosis of Crohn's Disease.
* IFX initiated as clinically indicated.
* Concurrent use of immunomodulators allowed.
* Endoscopy and/OR imaging depending on disease areas in the GI tract last 3 months (Paris classification/Simple Endoscopic Score - SES-CD).

Exclusion Criteria:

• Past exposure to anti-TNF therapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with Crohn's Disease whose treating physician has planned to start IFX for treatment of their CD.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The proportion of children with IFX trough level with the range of 5 to 10 µg/ml | at Week 10

SECONDARY OUTCOMES:
The proportion of children with IFX trough level within the range of 5 to 10 µg/ml | at week 14
  however, participants are being treated as per standard of care. It may be possible that the dose may be administered early as deemed necessary by treating provider.
Proportion in clinical remission and symptom response using the pediatric Crohn's disease activity index (PCDAI) | Beginning of the maintenance dose at the 5th dose of treatment/week 22
  This level will be measured prior to the 5th dose. Ideally, this will done at week 22; however, participants are being treated as per standard of care. It may be possible that the dose may be administered early as deemed necessary by treating provider.

CONTACTS AND LOCATIONS:
Overall Officials: Hien Q Huynh, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - SickKids, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Lamireau T, Cezard JP, Dabadie A, Goulet O, Lachaux A, Turck D, Maurage C, Morali A, Sokal E, Belli D, Stoller J, Cadranel S, Ginies JL, Viola S, Huet F, Languepin J, Lenaerts C, Bury F, Sarles J; French-Speaking Group for Pediatric Gastroenterology Nutrition. Efficacy and tolerance of infliximab in children and adolescents with Crohn's disease. Inflamm Bowel Dis. 2004 Nov;10(6):745-50. doi: 10.1097/00054725-200411000-00008. PMID 15626892
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Hyams J, Crandall W, Kugathasan S, Griffiths A, Olson A, Johanns J, Liu G, Travers S, Heuschkel R, Markowitz J, Cohen S, Winter H, Veereman-Wauters G, Ferry G, Baldassano R; REACH Study Group. Induction and maintenance infliximab therapy for the treatment of moderate-to-severe Crohn's disease in children. Gastroenterology. 2007 Mar;132(3):863-73; quiz 1165-6. doi: 10.1053/j.gastro.2006.12.003. Epub 2006 Dec 3. PMID 17324398
- [Background] Nanda KS, Cheifetz AS, Moss AC. Impact of antibodies to infliximab on clinical outcomes and serum infliximab levels in patients with inflammatory bowel disease (IBD): a meta-analysis. Am J Gastroenterol. 2013 Jan;108(1):40-7; quiz 48. doi: 10.1038/ajg.2012.363. Epub 2012 Nov 13. PMID 23147525
- [Background] Singh N, Rosenthal CJ, Melmed GY, Mirocha J, Farrior S, Callejas S, Tripuraneni B, Rabizadeh S, Dubinsky MC. Early infliximab trough levels are associated with persistent remission in pediatric patients with inflammatory bowel disease. Inflamm Bowel Dis. 2014 Oct;20(10):1708-13. doi: 10.1097/MIB.0000000000000137. PMID 25153505
- [Background] Maser EA, Villela R, Silverberg MS, Greenberg GR. Association of trough serum infliximab to clinical outcome after scheduled maintenance treatment for Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1248-54. doi: 10.1016/j.cgh.2006.06.025. Epub 2006 Aug 22. PMID 16931170
- [Background] Lamblin, C, Auburg,A, Ternant, D, Picon,L, Lecomte, T, and Paintaud, G. Concentration effect relationship of infliximab in Crohn's disease: Results of a cohort study. Journal of Crohn's and Colitis 2012; 6: S142-S143.
- [Background] Arias, MT, Vande, CN, Drobne, D et al. Importance of trough levels and antibodies on the long-term efficacy of infliximab therapy in ulcerative colitis. Journal of Crohn's and Colitis 2012; 6: s5.
- [Background] Wang SL, Ohrmund L, Hauenstein S, Salbato J, Reddy R, Monk P, Lockton S, Ling N, Singh S. Development and validation of a homogeneous mobility shift assay for the measurement of infliximab and antibodies-to-infliximab levels in patient serum. J Immunol Methods. 2012 Aug 31;382(1-2):177-88. doi: 10.1016/j.jim.2012.06.002. Epub 2012 Jun 9. PMID 22691619
- [Background] Hyams JS, Ferry GD, Mandel FS, Gryboski JD, Kibort PM, Kirschner BS, Griffiths AM, Katz AJ, Grand RJ, Boyle JT, et al. Development and validation of a pediatric Crohn's disease activity index. J Pediatr Gastroenterol Nutr. 1991 May;12(4):439-47. PMID 1678008
- [Background] Levine A, Griffiths A, Markowitz J, Wilson DC, Turner D, Russell RK, Fell J, Ruemmele FM, Walters T, Sherlock M, Dubinsky M, Hyams JS. Pediatric modification of the Montreal classification for inflammatory bowel disease: the Paris classification. Inflamm Bowel Dis. 2011 Jun;17(6):1314-21. doi: 10.1002/ibd.21493. Epub 2010 Nov 8. PMID 21560194
- See also: Study is being facilitated using the Canadian Children IBD Network — http://www.cidscann.ca/